CLINICAL TRIAL: NCT01130883
Title: Evaluation of Effectiveness of the Treatment After Repeated Administration of Klacid®SR in Patients With Upper Respiratory Infection, Exacerbation of Chronic Bronchitis and Mild Community-acquired Pneumonia in Common Clinical Practice in the Czech Republic
Brief Title: Evaluation of Effectiveness of the Treatment After Repeated Administration of Klacid®SR
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P12-109
Record Dates: First submitted 2010-05-06; First posted 2010-05-26 (Estimated); Results first posted 2011-08-23 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2011-09

CONDITIONS: Tracheitis; Tracheobronchitis; Bronchitis; Chronic Bronchitis; Community-Acquired Pneumonia (CAP)
Keywords: acute tracheitis; acute tracheobronchitis or acute bronchitis; acute exacerbation of chronic bronchitis; mild community-acquired pneumonia
MeSH Terms: conditions — Tracheitis; Bronchitis; Bronchitis, Chronic; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Respiratory Infections: Czech patients with acute tracheitis, acute tracheobronchitis or acute bronchitis; or patients with acute exacerbation of chronic bronchitis (AECB) or mild community-acquired pneumonia (CAP) who received Klacid®SR treatment 6 weeks prior to the next Klacid®SR dose or in intervals: 7-week - 3- month, 4- month - 12- month, 13- month - 24- month prior to the next Klacid®SR dose (next Klacid®SR dose = dose administered within this PMOS).

SUMMARY:
This post-marketing observational study (PMOS) will be conducted in a prospective, single-arm, single-country, multicenter format. The investigational sites will be consulting rooms of GPs (general practitioner), pneumologists and centers with experience in the treatment of patients with acute infections of trachea, bronchi, AECB (acute exacerbation of chronic bronchitis) and CAP (mild community-acquired pneumonia). Since this will be a post-marketing observational study, Klacid SR will be prescribed in usual manner in accordance with the terms of the local market authorization with regards to dose, population and indication as well as local guidelines. Objective: to describe the effectiveness of the treatment with repeated administration of Klacid SR in patients with acute tracheitis, acute tracheobronchitis or acute bronchitis; or in patients with acute exacerbation of chronic bronchitis (AECB) or mild community-acquired pneumonia (CAP) who received Klacid SR treatment 6 weeks to 24 months prior to the Klacid SR dose administered within this study.

DETAILED DESCRIPTION:
Follow-up of participants should enable three visits during this period. At the Screening Visit the decision for Klacid SR therapy in a dose of 500 -1000 mg once daily will be made. The Second Visit will occur 8 - 16 days after study initiation. The Last Visit will be a phone call to the participant after 30 days from the initiation of the treatment. Study visits will be defined as "V1" = Screening Visit, "V2" = Visit in which Klacid SR therapy will be terminated and "V3" = Phone call 30 days after initiation of Klacid SR therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men, women at least 18 years old.
* Patients treated with Klacid®SR between 6 weeks and 24 months prior to start of the PMOS.
* Patients:

  * with acute tracheitis,
  * acute tracheobronchitis,
  * acute bronchitis,
  * mild community-acquired pneumonia or
  * acute exacerbation of chronic bronchitis

Exclusion Criteria:

* Patients without previous administration of Klacid®SR and patients who used Klacid®SR less than 6 weeks ago or more than 24 months ago. The information about previous administration of Klacid®SR will be based on physician records or patients anamnesis.
* Patients with known hypersensitivity to macrolide antibiotics
* Patients with documented renal impairment (creatinine clearance under 30 ml/min).
* Patients with documented liver parenchyma impairment (AST, ALT and GMT > 3x higher level in comparison with the norm)
* Concomitant therapy with the following drugs: astemizole, cisapride, colchicine, pimozide, terfenadine and ergotamine or dihydroergotamine
* Pregnancy
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with: acute tracheitis, acute tracheobronchitis or acute bronchitis, acute exacerbation of chronic bronchitis, mild community-acquired pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 3130 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Hloska, M.D., Study Director — Abbott Laboratories, s.r.o. (Czech Republic)
Locations (135):
- Czechia (135):
  - Site Reference ID/Investigator# 37381, Bílina
  - Site Reference ID/Investigator# 37391, Bílina
  - Site Reference ID/Investigator# 37282, Blansko
  - Site Reference ID/Investigator# 37324, Blansko
  - Site Reference ID/Investigator# 37424, Boskovice
  - Site Reference ID/Investigator# 37329, Brandýs nad Labem
  - Site Reference ID/Investigator# 37268, Brno
  - Site Reference ID/Investigator# 37299, Brno
  - Site Reference ID/Investigator# 37331, Brno
  - Site Reference ID/Investigator# 37396, Brno
  - Site Reference ID/Investigator# 37411, Brno
  - Site Reference ID/Investigator# 37403, Brno
  - Site Reference ID/Investigator# 37380, Brno
  - Site Reference ID/Investigator# 37327, Brno
  - Site Reference ID/Investigator# 37443, Břeclav
  - Site Reference ID/Investigator# 37429, Bučovice
  - Site Reference ID/Investigator# 37444, Bučovice
  - Site Reference ID/Investigator# 37433, Buštěhrad
  - Site Reference ID/Investigator# 37362, Cheb
  - Site Reference ID/Investigator# 47286, Cheb
  - Site Reference ID/Investigator# 37413, Chrudim
  - Site Reference ID/Investigator# 37374, Čáslav
  - Site Reference ID/Investigator# 37267, České Budějovice
  - Site Reference ID/Investigator# 37269, České Budějovice
  - Site Reference ID/Investigator# 37298, České Budějovice
  - Site Reference ID/Investigator# 37302, České Budějovice
  - Site Reference ID/Investigator# 37392, České Budějovice
  - Site Reference ID/Investigator# 37408, České Budějovice
  - Site Reference ID/Investigator# 37372, Děčín
  - Site Reference ID/Investigator# 37394, Děčín
  - Site Reference ID/Investigator# 37263, Holešov
  - Site Reference ID/Investigator# 43230, Holešov
  - Site Reference ID/Investigator# 26623, Hradec Králové
  - Site Reference ID/Investigator# 37270, Hradec Králové
  - Site Reference ID/Investigator# 37371, Hradec Králové
  - Site Reference ID/Investigator# 43225, Hradec Králové
  - Site Reference ID/Investigator# 37367, Hranice
  - Site Reference ID/Investigator# 37274, Hrádek
  - Site Reference ID/Investigator# 37364, Hřebeč
  - Site Reference ID/Investigator# 37404, Jablonec nad Nisou
  - Site Reference ID/Investigator# 47283, Jablonec nad Nisou
  - Site Reference ID/Investigator# 43229, Jaroměř
  - Site Reference ID/Investigator# 37376, Jindřichův Hradec
  - Site Reference ID/Investigator# 37290, Kaplice
  - Site Reference ID/Investigator# 37369, Karlovy Vary
  - Site Reference ID/Investigator# 37445, Karlovy Vary
  - Site Reference ID/Investigator# 37363, Karlovy Vary
  - Site Reference ID/Investigator# 37283, Kladno
  - Site Reference ID/Investigator# 37382, Kolín
  - Site Reference ID/Investigator# 37368, Konice
  - Site Reference ID/Investigator# 37415, Konice
  - Site Reference ID/Investigator# 37272, Kralovice
  - Site Reference ID/Investigator# 42162, Kunovice
  - Site Reference ID/Investigator# 43224, Kyjov
  - Site Reference ID/Investigator# 37323, Letohrad
  - Site Reference ID/Investigator# 37389, Liberec
  - Site Reference ID/Investigator# 37416, Litomyšl
  - Site Reference ID/Investigator# 37384, Litvínov
  - Site Reference ID/Investigator# 37428, Mariánské Lázně
  - Site Reference ID/Investigator# 37289, Mělník
  - Site Reference ID/Investigator# 37293, Městec Králové
  - Site Reference ID/Investigator# 43228, Mohelnice
  - Site Reference ID/Investigator# 43233, Mohelnice
  - Site Reference ID/Investigator# 43227, Moravská Třebová
  - Site Reference ID/Investigator# 47290, Most
  - Site Reference ID/Investigator# 37297, Neratovice
  - Site Reference ID/Investigator# 37397, Nový Bor
  - Site Reference ID/Investigator# 37303, Nový Jičín
  - Site Reference ID/Investigator# 37400, Nový Jičín
  - Site Reference ID/Investigator# 37399, Obříství
  - Site Reference ID/Investigator# 37279, Olomouc
  - Site Reference ID/Investigator# 37280, Olomouc
  - Site Reference ID/Investigator# 37395, Pardubice
  - Site Reference ID/Investigator# 37271, Pilsen
  - Site Reference ID/Investigator# 37273, Pilsen
  - Site Reference ID/Investigator# 37423, Pilsen
  - Site Reference ID/Investigator# 37431, Pilsen
  - Site Reference ID/Investigator# 47284, Planá
  - Site Reference ID/Investigator# 37325, Poděbrady
  - Site Reference ID/Investigator# 47282, Poděbrady
  - Site Reference ID/Investigator# 37375, Prague
  - Site Reference ID/Investigator# 37398, Prague
  - Site Reference ID/Investigator# 37410, Prague
  - Site Reference ID/Investigator# 37387, Prague
  - Site Reference ID/Investigator# 37390, Prague
  - Site Reference ID/Investigator# 43232, Prague
  - Site Reference ID/Investigator# 43365, Prague
  - Site Reference ID/Investigator# 37288, Prague
  - Site Reference ID/Investigator# 37300, Prague
  - Site Reference ID/Investigator# 37301, Prague
  - Site Reference ID/Investigator# 37328, Prague
  - Site Reference ID/Investigator# 37330, Prague
  - Site Reference ID/Investigator# 37332, Prague
  - Site Reference ID/Investigator# 43236, Prague
  - Site Reference ID/Investigator# 37262, Prague
  - Site Reference ID/Investigator# 37295, Prague
  - Site Reference ID/Investigator# 37427, Prague
  - Site Reference ID/Investigator# 37275, Prague
  - Site Reference ID/Investigator# 37419, Prague
  - Site Reference ID/Investigator# 37438, Prague
  - Site Reference ID/Investigator# 37326, Prague
  - Site Reference ID/Investigator# 37414, Prague
  - Site Reference ID/Investigator# 47289, Prague
  - Site Reference ID/Investigator# 37291, Prague
  - Site Reference ID/Investigator# 37294, Prague
  - Site Reference ID/Investigator# 37437, Prostějov
  - Site Reference ID/Investigator# 37430, Prostějov
  - Site Reference ID/Investigator# 37378, Příbor
  - Site Reference ID/Investigator# 37412, Příbor
  - Site Reference ID/Investigator# 37432, Příbram
  - Site Reference ID/Investigator# 37425, Příbram
  - Site Reference ID/Investigator# 37442, Rakovník
  - Site Reference ID/Investigator# 37393, Raspenava
  - Site Reference ID/Investigator# 37421, Rožnov pod Radhoštěm
  - Site Reference ID/Investigator# 37287, Sadová
  - Site Reference ID/Investigator# 37406, Šlapanice
  - Site Reference ID/Investigator# 37383, Štětí
  - Site Reference ID/Investigator# 37278, Šumperk
  - Site Reference ID/Investigator# 43223, Šumperk
  - Site Reference ID/Investigator# 43234, Šumperk
  - Site Reference ID/Investigator# 37285, Tachov
  - Site Reference ID/Investigator# 37386, Teplice
  - Site Reference ID/Investigator# 37264, Třebíč
  - Site Reference ID/Investigator# 37277, Třebíč
  - Site Reference ID/Investigator# 43231, Třeboň
  - Site Reference ID/Investigator# 37405, Třinec
  - Site Reference ID/Investigator# 43366, Týn
  - Site Reference ID/Investigator# 37265, Týn nad Vltavou
  - Site Reference ID/Investigator# 37434, Uherské Hradiště
  - Site Reference ID/Investigator# 37365, Uherský Brod
  - Site Reference ID/Investigator# 37284, Velké Pavlovice
  - Site Reference ID/Investigator# 37385, Vlašim
  - Site Reference ID/Investigator# 37366, Zdar
  - Site Reference ID/Investigator# 43235, Zlín
  - Site Reference ID/Investigator# 37322, Žamberk

RESULTS

PARTICIPANT FLOW:
Groups:
- Klacid SR Treatment: Adult Czech participants with acute tracheitis, acute tracheobronchitis or acute bronchitis; or participants with acute exacerbation of chronic bronchitis (AECB) or mild community-acquired pneumonia (CAP) who received Klacid SR treatment 6 weeks to 24 months prior to the Klacid SR dose dose administered within this study.
Period: Overall Study
Arm/Group | Klacid SR Treatment
Started | 3130
Participants Analyzed | 3128
Completed | 3120
Not Completed | 10
Not completed — Patient Noncompliance | 6
Not completed — Reason Unknown | 1
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Klacid SR Treatment
Number analyzed (Participants) | 3130
Age, Customized [Number; unit: participants]
  less than 18 years of age | 2
  18 to 29 years of age | 281
  30 to 39 years of age | 544
  40 to 49 years of age | 589
  50 to 59 years of age | 680
  60 to 69 years of age | 630
  70 to 79 years of age | 305
  80 to 89 years of age | 92
  90 years of age and older | 7
Sex/Gender, Customized [Number; unit: Participants] — Gender was not reported in this study.
  Participants | 3130
Region of Enrollment [Number; unit: participants]
  Czech Republic | 3130

OUTCOME MEASURES:

1. Primary Outcome: Disappearance or Significant Alleviation of Symptoms
Description: Overall therapeutic response, "yes" or "no" was determined by the physician based on subjective response regarding disappearance or significant alleviation of symptoms following treatment. The physician also considered objective findings such as auscultation and or chest X-ray results (if available) when determining overall therapeutic response.
Time Frame: Day 8 - 16
Population: A total of 3130 participants were enrolled into the study and 3128 were included in the analysis. Two participants were excluded from the analysis as they did not meet entry criteria (2 participants were less than 18 years of age).
Measure: Number; unit: Participants
Arm/Group | Klacid SR Treatment
Number analyzed (Participants) | 3128
Participants | 3109

2. Primary Outcome: Change in Auscultation Findings, Regression of Chest X-ray Findings (Recorded by the Physician)
Description: Auscultation findings (abnormal breath sounds) were assessed at the initial visit (Day 0) and the second visit (Day 8 -16) by the physician. "Regression of chest X-ray findings" were not recorded as it is not part of routine clinical practice to confirm X-ray regression after the participant has clinically recovered from Community-Acquired Pneumonia (CAP).
Time Frame: Day 0, Day 8 - 16
Measure: Number; unit: participants
Arm/Group | Klacid SR Treatment
Number analyzed (Participants) | 3128
participants
  Initial Visit - Auscultation Normal | 956
  Initial Visit - Auscultation Abnormal | 2146
  Initial Visit - Findings Not Reported | 26
  Second Visit - Auscultation Normal | 2768
  Second Visit - Auscultation Abnormal | 247
  Second Visit - Findings Not Reported | 113

3. Secondary Outcome: Body Temperature
Description: Number of participants in which body temperature was increased (temperature above 37 degrees Celsius).
Time Frame: Day 0, Day 8-16
Population: Of the 3128 participants included in the analysis, body temperature was not reported for 6 participants at the Initial visit, and 14 participants at the Second visit.
Measure: Number; unit: Participants
Arm/Group | Klacid SR Treatment
Number analyzed (Participants) | 3128
Participants
  Initial Visit - Temperature above 37 degrees C | 2252
  Initial Visit - Temperature not above 37 degrees C | 870
  Initial Visit - Temperature not reported | 6
  Second Visit - Temperature above 37 degrees C | 101
  Second Visit - Temperature not above 37 degrees C | 3013
  Second Visit - Temperature not reported | 14

4. Secondary Outcome: Bacteriological Investigation (if Available)
Description: The type of agent present in the infection was assessed using bacteriological investigation. Occurrence of the most common agents was reported. Participants may have had more than one pathogen present. Test results were not available prior to enrollment but were reported during the study.
Time Frame: Day 0
Population: Of the 3128 participants included in the analysis, 225 participants had bacteriological investigations conducted at the Initial visit (Day 0). Some participants had more than one finding.
Measure: Number; unit: participants
Arm/Group | Klacid SR Treatment
Number analyzed (Participants) | 225
participants
  Haemophilus Influenzae | 48
  Streptococcus pneumoniae | 38
  Chlamydia pneumoniae | 34
  Mycoplasma pneumoniae | 14
  Haemophilus parainfluenzae | 13
  Klebsiella pneumoniae | 12
  Haemophilus species | 10
  Staphylococcus aureus | 5
  Branhamella catarrhalis | 5

5. Secondary Outcome: Cough and Its Character
Description: Number of participants in which cough was present, and if present, type of cough (irritating, productive, both or not reported)
Time Frame: Day 0, Day 8-16
Measure: Count of Participants; unit: Participants
Arm/Group | Klacid SR Treatment
Number analyzed (Participants) | 3128
Participants
  Initial Visit - Presence of cough | 2942
  a) Irritating cough | 1601
  b) Productive cough | 1177
  c) Both irritating and productive | 157
  d) Not Reported | 7
  Initial Visit -Cough not present | 186
  Second Visit -Presence of cough | 556
  a) Irritating cough. | 187
  b) Productive cough. | 351
  c) Both irritating and productive. | 16
  d) Not Reported. | 2
  Second Visit -Cough not present | 2572

6. Secondary Outcome: Dyspnea and Its Type
Description: Presence of dyspnea (difficulty breathing) and type of dyspnea (exertional, resting, both, or not reported).
Time Frame: Day 0, Day 8-16
Measure: Number; unit: Participants
Arm/Group | Klacid SR Treatment
Number analyzed (Participants) | 3128
Participants
  Initial Visit - Presence of dyspnea | 1091
  a) Exertional | 794
  b) Resting | 235
  c) Both exertional and resting | 60
  d) Type of dyspnea not reported | 2
  Initial Visit - Dyspnea not present | 2037
  Second Visit - Presence of dyspnea | 262
  a) Exertional- | 234
  b) Resting- | 17
  c) Both exertional and resting- | 9
  d) Type of dyspnea not reported- | 2
  Second Visit -Dyspnea not present | 2866

7. Secondary Outcome: Auscultation
Description: Participants with abnormal auscultation findings (abnormal breath sounds) and type of findings (wheezing, crackles, both, or not reported).
Time Frame: Day 0, Day 8-16
Population: Of the 3128 participants included in the analysis, auscultation findings were not reported for 38 participants at the initial visit and 116 participants at the final visit.
Measure: Number; unit: Participants
Arm/Group | Klacid SR Treatment
Number analyzed (Participants) | 3128
Participants
  Initial Visit - Abnormal Auscultaton findings | 2146
  a) Wheezing | 1577
  b) Crackles | 408
  c) Both wheezing and crackles | 145
  d) Not reported | 16
  Second Visit -Abnormal Auscultation findings | 247
  a) Wheezing- | 187
  b) Crackles- | 54
  c) Both wheezing and crackles- | 4
  d) Not reported- | 2

8. Secondary Outcome: Chest X-ray in Case of Community-Acquired Pneumonia (CAP)
Description: Number of participants in which X-ray findings were suggestive of pneumonia. In participants where the physician suspected CAP, a chest X-ray was performed and reviewed to determine whether findings were indicative of pneumonia.
Time Frame: Day 0
Population: Chest X-ray was performed in 294 of the participants for whom the physician suspected pneumonia.
Measure: Number; unit: Participants
Arm/Group | Klacid SR Treatment
Number analyzed (Participants) | 294
Participants
  Findings indicative of pneumonia | 276
  Findings not indicative of pneumonia | 18

9. Secondary Outcome: Study Drug Given as the First, Second or Third Antimicrobial Treatment
Description: Number of participants who received Klacid SR as the first, second or third (further) antimicrobial agent.
Time Frame: Day 0
Measure: Number; unit: Participants
Arm/Group | Klacid SR Treatment
Number analyzed (Participants) | 3128
Participants
  Klacid SR as first antimicrobial treatment | 2910
  Klacid SR as second antimicrobial treatment | 216
  Klacid SR as third antimicrobial treatment | 2

10. Secondary Outcome: Compliance
Description: Number of participants who took their medication according to the prescribed regimen (dose and duration) during the study.
Time Frame: Day 8 - 16
Measure: Number; unit: Participants
Arm/Group | Klacid SR Treatment
Number analyzed (Participants) | 3128
Participants | 3122

11. Secondary Outcome: Termination of Treatment Due to Noncompliance
Description: Number of participants who discontinued Klacid SR treatment early due to noncompliance with the recommended study medication regimen.
Time Frame: Day 8 - 16
Population: A total of 3128 participants were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Klacid SR Treatment
Number analyzed (Participants) | 3128
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the start to the completion of treatment with Klacid SR (8 to 16 days). Serious adverse events and relapse were reported for up to 30 days after the initiation of physician prescribed study treatment.
Description: Investigator monitored study participants for adverse events as per usual practice.
Arm/Group | Klacid SR Treatment
Serious Adverse Events (participants affected / at risk) | 2/3128
Other Adverse Events (participants affected / at risk) | 7/3128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Klacid SR Treatment (N=3128)
Tuberculosis pleuritis (Infections and infestations) | 1
Pulmonary tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Klacid SR Treatment (N=3128)
Bad taste in mouth (Gastrointestinal disorders) | 1
Loss of appetite (General disorders) | 1
Burning tongue (Gastrointestinal disorders) | 1
Bitter taste in mouth (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Gastrointestinal tract symptoms (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.